CLINICAL TRIAL: NCT01041066
Title: Nicardipine Versus Labetalol During Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Seoul National University Bundang Hospital, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: nicardipine-labetalol
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2009-12-31 (Estimated); Status verified 2009-09

CONDITIONS: Patients Who Are Intubated for General Anesthesia; Endotracheal Intubation
Keywords: patients who are intubated for general anesthesia
MeSH Terms: interventions — Labetalol; Nicardipine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- group L (Active Comparator): 0.4 mg/kg labetalol
  Interventions: Drug: labetalol
- group N (Active Comparator): 20 ㎍/kg nicardipine
  Interventions: Drug: nicardipine

INTERVENTIONS:
Drug: labetalol — 0.4 mg/kg labetalol intravenously 4 min before intubation
  Arms: group L
Drug: nicardipine — 20 ㎍/kg nicardipine intravenously 4 min before intubation
  Arms: group N

SUMMARY:
The aim of this study was to compare the efficacy of nicardipine and labetalol in attenuation of cardiovascular responses to endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for general anesthesia with endotracheal intubation

Exclusion Criteria:

* Patients with heart failure or coronary artery disease 2-3 degree atrio-ventricular block or severe bradycardia (< 45 beats/min) asthma, bronchial spasm or chronic obstructive pulmonary disease patients with anticipated difficult intubation (Mallampati class III, IV) severe hepatic or renal dysfunction allergy or contraindication to study medication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
hemodynamic variables (systolic blood pressure, diastolic blood pressure and mean blood pressure, heart rate) | preinduction- 10 min after intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Ryu JH, Apfel CC, Whelan R, Jeon YT, Hwang JW, Do SH, Ro YJ, Kim CS. Comparative prophylactic and therapeutic effects of intravenous labetalol 0.4 mg/kg and nicardipine 20 mug/kg on hypertensive responses to endotracheal intubation in patients undergoing elective surgeries with general anesthesia: a prospective, randomized, double-blind study. Clin Ther. 2012 Mar;34(3):593-604. doi: 10.1016/j.clinthera.2012.01.017. Epub 2012 Feb 24. PMID 22364823